CLINICAL TRIAL: NCT06868277
Title: A Phase III, Randomized, Double-blind, Multicenter, Global Study of Rilvegostomig or Pembrolizumab Monotherapy for the First-line Treatment of Patients With PD-L1-high Metastatic Non-small Cell Lung Cancer (ARTEMIDE-Lung04)
Brief Title: A Global Phase III Study of Rilvegostomig or Pembrolizumab Monotherapy for First-Line Treatment of PD-L1-high Metastatic Non-small Cell Lung Cancer
Acronym: ARTEMIDELung04
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D702GC00001; 2024-517780-24-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: ARTEMIDE-Lung04; Rilvegostomig (AZD2936); Non-small cell lung cancer (NSCLC); Bi-specific antibody; T-cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif domain (TIGIT); EGFR, ALK and ROS1 testing; Programmed cell death protein (PD-L1); Pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to one of the following intervention arms:
  Arm A : Rilvegostomig Arm B : Pembrolizumab
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Drug: rilvegostomig
  Interventions: Biological: Rilvegostomig
- Arm B (Active Comparator): Drug: Pembrolizumab
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Rilvegostomig — Administered intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: AZD2936
  Arms: Arm A
Biological: Pembrolizumab — Administered intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: KEYTRUDA
  Arms: Arm B

SUMMARY:
The purpose of ARTEMIDE-Lung04 is to assess the efficacy and safety of rilvegostomig compared with pembrolizumab monotherapy as 1L treatment in participants with mNSCLC and whose tumors express PD-L1.

DETAILED DESCRIPTION:
This is a Phase III, two-arm, randomized, double-blind, global, multicenter study assessing the efficacy and safety of rilvegostomig compared to pembrolizumab as a 1L treatment for patients with mNSCLC whose tumors express PD-L1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented NSCLC (non small lung cancer), including all histological subtypes.
* Stage IV mNSCLC (metastatic non-small cell lung cancer) (based on the American Joint Committee on Cancer Edition 8) not amenable to curative treatment.
* Absence of sensitizing EGFR (epidermal growth factor) mutations and ALK (anaplastic lymphoma kinase) and ROS1 (c-ros oncogene 1) rearrangements. Negative assay result is required for all non-squamous histology subtypes.
* Absence of documented tumor genomic mutation results from tests conducted as part of standard local practice in any other actionable driver oncogenes for which there are locally approved targeted 1L (first line) therapies.
* WHO (World Health Organization)/ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1, with no deterioration over the previous 2 weeks prior to baseline at screening and prior to randomization.
* Minimum life expectancy of 12 weeks.
* Provision of acceptable tumor sample for the central testing prior to randomization.
* At least one lesion not previously irradiated that qualifies as a RECIST 1.1 (Response Evaluation Criteria in Solid Tumors, Version 1.1) TL (target lesion) at baseline and can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with CT (computed tomography) or MRI (magnetic resonance imaging) and is suitable for accurate repeated measurements.
* Adequate organ and bone marrow function

Exclusion Criteria:

* As judged by the investigator, any severe or uncontrolled systemic diseases, makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.
* History of organ transplant.
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence.
* Presence of small cell and neuroendocrine histology components.
* Brain metastases unless asymptomatic, stable, and not requiring steroids or anticonvulsants for at least 4 weeks prior to start of study intervention.
* Active primary immunodeficiency/active infectious disease(s)
* Active tuberculosis infection
* Any prior systemic therapy received for advanced or mNSCLC (metastatic non-small cell lung cancer).
* Any prior exposure to an anti-TIGIT (T-cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif domain) therapy or any other anticancer therapy targeting immune-regulatory receptors or mechanisms.
* Any prior treatment with an anti-PD-1 (programmed cell death protein 1) or anti-PD-L1 (anti-programmed death-ligand 1) agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2030-01-17 (Estimated); Study Completion 2030-12-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization until the date of death due to any cause.
Progression-Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1 or death due to any cause (in the absence of progression).

SECONDARY OUTCOMES:
Landmark Overall Survival (OS) rates | Up to approximately 5 years
  OS is defined as the time from randomization until the date of death due to any cause.
Landmark Progression-Free Survival (PFS) rates | Up to approximately 5 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1 or death due to any cause (in the absence of progression).
Objective Response Rate (ORR) | Up to approximately 5 years
  ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR, using RECIST 1.1.
Duration of Response (DoR) | Up to approximately 5 years
  DoR is defined as the time from the date of first documented response until the date of documented progression using RECIST 1.1 or death due to any cause (in the absence of progression).
Time to second progression or death (PFS2) | Up to approximately 5 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial investigator-assessed progression event), after the start of the first subsequent therapy, or death from any cause, whichever occurs first.
Pharmakokinetics (PK) of rilvegostomig | Up to approximately 5 years
  Concentration of rilvegostomig in serum
Immunogenicity of rilvegostomig | Up to approximately 5 years
  Presence of antidrug antibodies (ADAs), titer, and neutralizing antibodies for rilvegostomig.
Patient-reported physical functioning | Up to approximately 5 years
  Proportion of participants with maintained or improved physical functioning as measured by Patient-Reported Outcomes Measurement Information System Physical Function - Short Form 8c - 7 day (PROMIS PF-SF 8c - 7 day) at each time point.
Patient-reported global health status (GHS)/quality of life (QoL) | Up to approximately 5 years
  Time to deterioration (TTD) of GHS/QoL as measured by the European Organization for Research and Treatment of Cancer Item Library 172 (EORTC IL172). TTD is defined as time from randomization to the date of first deterioration.
Patient-reported lung cancer symptoms of non-small cell lung cancer (NSCLC) | Up to approximately 5 years
  Time to deterioration (TTD) in pulmonary symptoms as measured by the Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ).
  TTD is defined as time from randomization to the date of first deterioration.

CONTACTS AND LOCATIONS:
Locations (232):
- United States (29):
  - Research Site, Bay Pines, Florida
  - Research Site, Clearwater, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Des Moines, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Leawood, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Bridgeton, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Paramus, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, East Syracuse, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, Westbury, New York
  - Research Site, Canton, Ohio
  - Research Site, Fountain Hill, Pennsylvania
  - Research Site, Kittanning, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Round Rock, Texas
  - Research Site, Aberdeen, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Morgantown, West Virginia
- Argentina (4):
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, Rosario
  - Research Site, Viedma
- Australia (2):
  - Research Site, Hobart
  - Research Site, Woolloongabba
- Belgium (6):
  - Research Site, Edegem
  - Research Site, Jette
  - Research Site, Libramont-Chevigny
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Roeselaere
- Brazil (12):
  - Research Site, Blumenau
  - Research Site, Fortaleza
  - Research Site, Ijuí
  - Research Site, Itajaí
  - Research Site, Londrina
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Porto Velho
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Teresina
- Bulgaria (4):
  - Research Site, Burgas
  - Research Site, Panagyurishte
  - Research Site, Sofia
  - Research Site, Varna
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Cambridge, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saint-Jérôme, Quebec
- Chile (2):
  - Research Site, Conception
  - Research Site, Santiago
- China (30):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haerbin
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jiamusi
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Liuchow
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Xuzhou
  - Research Site, Yantai
  - Research Site, Zhengzhou
- Colombia (4):
  - Research Site, Cali
  - Research Site, Floridablanca
  - Research Site, Medellín
  - Research Site, Valledupar
- Costa Rica (2):
  - Research Site, San José
  - Research Site, Santa Ana
- France (13):
  - Research Site, Angers
  - Research Site, Avignon
  - Research Site, Boulogne-Billancourt
  - Research Site, Caen
  - Research Site, Chambéry
  - Research Site, Dijon
  - Research Site, La Tronche
  - Research Site, Limoges
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, St-Malo
  - Research Site, Toulouse
- Research Site, Tbilisi, Georgia
- Germany (23):
  - Research Site, Amberg
  - Research Site, Augsburg, by
  - Research Site, Bad Saarow
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Braunschweig
  - Research Site, Essen
  - Research Site, Flensburg
  - Research Site, Frankfurt am Main
  - Research Site, Heilbronn
  - Research Site, Immenhausen
  - Research Site, Koblenz
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Oldenburg
  - Research Site, Rotenburg (Wümme)
  - Research Site, Schweinfurt
  - Research Site, Trier
  - Research Site, Velbert
  - Research Site, Wuppertal
  - Research Site, Würselen
  - Research Site, Würzburg
- Greece (3):
  - Research Site, Athens
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Ireland (2):
  - Research Site, Dublin
  - Research Site, Galway
- Israel (7):
  - Research Site, Afula
  - Research Site, Beersheba
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (11):
  - Research Site, Candiolo
  - Research Site, Lecco
  - Research Site, Lucca
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Peschiera del Garda
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Udine
  - Research Site, Verona
- Japan (23):
  - Research Site, Akashi
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Iwakuni-shi
  - Research Site, Izumi-shi
  - Research Site, Kashihara-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nankoku-shi
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Takarazuka-shi
  - Research Site, Toon-Shi
  - Research Site, Toyoake-shi
  - Research Site, Toyonaka-shi
- Malaysia (5):
  - Research Site, George Town
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Perai
- Portugal (7):
  - Research Site, Alcabideche
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
- Romania (7):
  - Research Site, Bucharest
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Otopeni
  - Research Site, Piteşti
  - Research Site, Sibiu
  - Research Site, Timișoara
- South Korea (2):
  - Research Site, Jinju
  - Research Site, Seoul
- Spain (14):
  - Research Site, Badajoz
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Granada
  - Research Site, Jaén
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Valencia
  - Research Site, Vigo (Pontevedra)
  - Research Site, Zaragoza
- Research Site, Lausanne, Switzerland
- Turkey (Türkiye) (6):
  - Research Site, Ankara
  - Research Site, Bakırköy
  - Research Site, Çankaya
  - Research Site, İzmit
  - Research Site, Küçükçekmece
  - Research Site, Yüreğir
- United Kingdom (5):
  - Research Site, Blackpool
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, Hull
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/